CLINICAL TRIAL: NCT04906317
Title: The Effectiveness of Sedation and Analgesia in Colonoscopy Treatment of Colorectal Polyps: a Single-center, Prospective, Randomized Controlled Study
Brief Title: The Effectiveness of Sedation and Analgesia in Colonoscopy Treatment of Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021ZSLYEC-028
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Colonoscopy; Sedation and Analgesia
MeSH Terms: conditions — Agnosia | interventions — Midazolam; dezocine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation and Analgesia (Active Comparator): 0.05 mg/kg midazolam and 5mg dezocine iv infusion
  Interventions: Drug: midazolam and dezocine
- Anesthesia (Active Comparator): continuous 1.5mg/kg propofol iv infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: midazolam and dezocine — Midazolam (0.05 mg/kg) and dezocine(5mg) sedation during colonoscopy, targeted to a painless level
  Other Names: Not necessary
  Arms: Sedation and Analgesia
Drug: Propofol — standard propofol (1.5mg/kg) induction during colonoscopy, targeted to a moderate sedation level
  Other Names: Not necessary
  Arms: Anesthesia

SUMMARY:
This study aims to evaluate the effectiveness of sedation and analgesia in the treament of colorectal polyps by colonoscopy.

DETAILED DESCRIPTION:
Colorectal polyps are precancerous lesions of the colorectal cancer. Colonoscopy can reduce the risk of colorectal cancer. Painless endoscopy could reduce patient discomfort and improves the acceptance of treatment, especially for the endoscopic treatment of colorectal polyps. Intravenous anesthesia colonoscopy has a strong sedative effect and has obvious inhibitory effects on the respiratory and circulatory systems. It requires the assistance of an anesthesiologist. The lack of anesthesiologists makes it difficult to make an appointment for anesthesia colonoscopy, which is a bottleneck in the diagnosis and treatment of gastrointestinal diseases in China. Therefore, there is an urgent need to find a painless diagnosis and treatment method that is not inferior to anesthesia colonoscopy in comfort to meet the needs of patients. Comparing to anesthesia colonoscopy, sedative and analgesic colonoscopy have similar sedative and analgesic effects and do not require the assistance of an anesthesiologist. However, there is no relevant evaluation on the effectiveness of sedation and analgesia during the endoscopic treatment of colorectal polyps. Our department has used midazolam combined with dezocine to treat 185 patients with colorectal polyps in these years. Retrospective analysis showed that the sedative and analgesic effect is satisfactory. Therefore, it is necessary to make a single-center randomized parallel group controlled non-inferiority study to directly compare the effectiveness of sedation and analgesia versus intravenous anesthesia in endoscopic treatment of colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy diagnosed as a colorectal polyp, the number of polyps is less than 5, and the size of single polyp is less than 2.0 cm
* Age more than 18 years and less than 70 years

Exclusion Criteria:

* Allergy to propofol, dezocine, midazolam or eggs
* ASA class IV, short and tick neck, difficult intubation due to inability to open the mouth widely
* Suspected of gastrointestinal perforation, bleeding or obstruction
* Acute gastrointestinal infection period
* History of abdominal surgery
* Patients during pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
The score of visual analogue scoring (VAS) | immediately after the procedure of colonoscopy
  Assess immediately after the completement of colonoscopy

SECONDARY OUTCOMES:
Treatment fee | During the colonoscopy procedure
  The fee of treatment refers to the total cost of anesthesia fee, anesthesia/sedation drug fee, intraoperative monitoring fee, endoscopy fee and endoscopic treatment fee

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Guo, MD, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Six Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No